CLINICAL TRIAL: NCT01716806
Title: A Phase 2 Open-label Study of Brentuximab Vedotin in Front-line Therapy of Hodgkin Lymphoma (HL) an dCD30-expressing Peripheral T-cell Lymphoma (PTCL) in Older Patients or Patients With Significant Comorbidities Ineligible for Standard Chemotherapy
Brief Title: A Study of Brentuximab Vedotin With Hodgkin Lymphoma (HL) and CD30-expressing Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-015
Record Dates: First submitted 2012-10-16; First posted 2012-10-30 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Hodgkin Disease; Peripheral T Cell Lymphoma
Keywords: Antibody-Drug Conjugate; Antibodies, Monoclonal; Hematologic Diseases; Hodgkin Disease; Antigens, CD30; Lymphoma; monomethylauristatin E; Drug Therapy; CD30-expression; PTCL; Seattle Genetics
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Bendamustine Hydrochloride; Dacarbazine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: Brentuximab Vedotin in HL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin
- Part B: Brentuximab Vedotin + Dacarbazine in HL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin; Drug: dacarbazine
- Part C: Brentuximab Vedotin + Bendamustine in HL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin; Drug: bendamustine
- Part D: Brentuximab Vedotin + Nivolumab in HL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin; Drug: nivolumab
- Part E: Brentuximab Vedotin in HL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin
- Part F: Brentuximab Vedotin in PTCL Patients (Experimental)
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by IV infusion
  Other Names: Adcetris; SGN-35
Drug: bendamustine — 70 mg/m^2 by IV infusion on Days 1 and 2 of 3-week cycle
  Arms: Part C: Brentuximab Vedotin + Bendamustine in HL Patients
Drug: dacarbazine — 375 mg/m^2 every 3 weeks by IV infusion
  Arms: Part B: Brentuximab Vedotin + Dacarbazine in HL Patients
Drug: nivolumab — 3 mg/kg every 3 weeks by IV infusion
  Arms: Part D: Brentuximab Vedotin + Nivolumab in HL Patients

SUMMARY:
This trial will study brentuximab vedotin to find out whether it is an effective treatment for Hodgkin lymphoma (HL) and peripheral T-cell lymphoma (PTCL). Participants in this study will be older or will have other conditions that make them unable to have standard chemotherapy treatment. The study will look at brentuximab vedotin alone and combined with other drugs.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and tolerability of brentuximab vedotin as monotherapy and in combination with other agents as frontline therapy. There are 6 parts of the study. The population to be studied includes treatment-naïve patients with classical Hodgkin lymphoma (HL) or treatment-naïve patients with CD30-expressing peripheral T-cell lymphoma (PTCL).

ELIGIBILITY:
Inclusion Criteria:

* Parts A, B, C, and D: 60 years of age or older
* Treatment-naive patients with histopathological diagnosis of classical Hodgkin lymphoma (Parts A, B, C, D, and E)
* Treatment-naive patients with CD30-expressing PTCL (Part F)
* Ineligible for or have declined initial conventional combination chemotherapy for HL (Parts A, B, C, and D)
* Unsuitable or unfit for initial conventional combination chemotherapy for HL (Part E) or CD30-expressing PTCL due to the presence of comorbidity-factors, as documented by:

  * A CIRS score of 10 or greater
  * Requiring assistance with or dependence on other for any instrumental activities of daily living (IADLs)
* Measurable disease of at least 1.5 cm as documented by radiographic technique
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 3 (Parts, A, B, C, E, and F) or less than or equal to 2 (Part D)

Exclusion Criteria:

* Symptomatic neurologic disease compromising IADLs or requiring medication
* History of progressive multifocal leukoencephalopathy
* Grade 3 or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of brentuximab vedotin
* Concurrent use of other investigational agents
* Chemotherapy, radiotherapy, biologics, and/or other treatment with immunotherapy not completed 4 weeks prior to first dose of study drug
* History of another malignancy within 1 year before first dose of study drug (Parts E and F only)
* Part D only:

  * Received any prior immune-oncology therapy
  * History of known or suspected autoimmune disease
  * Prior allogeneic stem cell transplant
  * History of cerebral vascular event within 6 months of first dose of study drug
  * Active interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicology
  * Known history of pancreatitis
* Parts D, E, and F only:

  * Known cerebral/meningeal disease related to the underlying malignancy
  * Systemic treatment with corticosteroids or other immunosuppressive medications within 1 week of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sims, MD, Study Director — Seagen Inc.
Locations (54):
- United States (49):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama - Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Urological Institute, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Arizona Cancer Center / University of Arizona, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Providence St Joseph Medical Center, Burbank, California
  - City of Hope National Medical Center, Duarte, California
  - Wilshire Oncology Medical Group Inc., Pomona, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Florida Cancer Affiliates, Trinity, Florida
  - IACT Health, Columbus, Georgia
  - Georgia Cancer Specialists / Northside Hospital Cancer Institute, Sandy Springs, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Specialists / Advocate Lutheran General Hospital, Niles, Illinois
  - American Oncology Networks LLC, Bethesda, Maryland
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Minnesota Oncology Hematology P.A., Minneapolis, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Morristown Medical Center/ Carol G. Simon Cancer Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Prisma Health, Greenville, South Carolina
  - Arlington Cancer Center, Arlington, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology - Fort Worth 12th Avenue, Fort Worth, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Oncology - Longview, Longview, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Seton Williamson, Round Rock, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Oncology and Hematology Assoc of SW VA DBA Blue Ridge Cancer Care, Salem, Virginia
  - Shenandoah Oncology P.C., Winchester, Virginia
  - Benaroya Research Institute/Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - University of Alberta / Cross Cancer Institute, Edmonton, Alberta
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - CIUSSS de L'Est de l'lle de Montreal / installation Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Friedberg JW, Bordoni R, Patel-Donnelly D, Larson T, Goldschmidt J, Boccia R, Cline VJM, Mamidipalli A, Liu J, Akyol A, Yasenchak CA. Brentuximab vedotin with dacarbazine or nivolumab as frontline cHL therapy for older patients ineligible for chemotherapy. Blood. 2024 Feb 29;143(9):786-795. doi: 10.1182/blood.2022019536. PMID 37946283
- [Derived] Friedberg JW, Forero-Torres A, Bordoni RE, Cline VJM, Patel Donnelly D, Flynn PJ, Olsen G, Chen R, Fong A, Wang Y, Yasenchak CA. Frontline brentuximab vedotin in combination with dacarbazine or bendamustine in patients aged >/=60 years with HL. Blood. 2017 Dec 28;130(26):2829-2837. doi: 10.1182/blood-2017-06-787200. Epub 2017 Oct 16. PMID 29038340
- [Derived] Forero-Torres A, Holkova B, Goldschmidt J, Chen R, Olsen G, Boccia RV, Bordoni RE, Friedberg JW, Sharman JP, Palanca-Wessels MC, Wang Y, Yasenchak CA. Phase 2 study of frontline brentuximab vedotin monotherapy in Hodgkin lymphoma patients aged 60 years and older. Blood. 2015 Dec 24;126(26):2798-804. doi: 10.1182/blood-2015-06-644336. Epub 2015 Sep 16. PMID 26377597
- [Derived] Gopal AK, Bartlett NL, Forero-Torres A, Younes A, Chen R, Friedberg JW, Matous JV, Shustov AR, Smith SE, Zain J, O'Meara MM, Fanale MA. Brentuximab vedotin in patients aged 60 years or older with relapsed or refractory CD30-positive lymphomas: a retrospective evaluation of safety and efficacy. Leuk Lymphoma. 2014 Oct;55(10):2328-34. doi: 10.3109/10428194.2013.876496. Epub 2014 Feb 24. PMID 24359243

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Brentuximab vedotin (BV) monotherapy in adults age 60 and above with classical Hodgkin Lymphoma (cHL). BV (1.8 mg/kg) was administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle.
- Part B: BV in combination with dacarbazine as frontline therapy in adults aged 60 and above with cHL. BV (1.8 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle. Dacarbazine (375 mg/m^2) was administered as an IV infusion on Day 1 of each 21-day cycle.
- Part C: BV in combination with bendamustine as frontline therapy in adults aged 60 and above with cHL. BV (1.8 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle. Bendamustine (70 mg/m^2) was administered as an IV infusion on Day 1 and Day 2 of each 21-day cycle.
- Part D: BV in combination with nivolumab as frontline therapy in adults aged 60 and above with cHL. BV (1.8 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle. Nivolumab (3 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle.
- Part E: BV as frontline monotherapy in patients with cHL who were unsuitable or unfit for combination chemotherapy. BV (1.8 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle.
- Part F: BV as frontline monotherapy in patients with CD30-expressing PTCL who were unsuitable or unfit for combination chemotherapy. BV (1.8 mg/kg) was administered as an IV infusion on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Started | 28 | 22 | 22 | 21 | 31 | 7
Received at Least One Dose of Study Drug | 27 | 22 | 20 | 21 | 30 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 28 | 22 | 22 | 21 | 31 | 7
Not completed — Patient withdrawal of consent | 4 | 2 | 4 | 3 | 2 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0 | 2 | 1 | 0
Not completed — Death | 13 | 9 | 12 | 4 | 10 | 5
Not completed — Received treatment past data cutoff of up to 16 doses of BV. AEs collected until end of study. | 0 | 0 | 0 | 0 | 1 | 1
Not completed — PI decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Change in performance status | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor terminated enrollment into Part C | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor direction | 7 | 8 | 5 | 12 | 16 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all participants who received any amount of brentuximab vedotin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F | Total
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 4 | 1 | 1 | 12
  >=65 years | 25 | 19 | 19 | 17 | 29 | 6 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 10 | 6 | 16 | 2 | 53
  Male | 14 | 16 | 10 | 15 | 14 | 5 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 0 | 1 | 2 | 2 | 11
  Not Hispanic or Latino | 25 | 18 | 20 | 20 | 28 | 5 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 2 | 0 | 0 | 6
  White | 26 | 19 | 20 | 19 | 26 | 7 | 117
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 0 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity, 1=Symptoms but ambulatory, 2=In bed <50% of the time, 3=In bed >50% of the time, 4=100% bedridden, 5=Dead
  Participants
    Grade 0 | 9 | 6 | 4 | 4 | 5 | 0 | 28
    Grade 1 | 12 | 9 | 12 | 16 | 10 | 4 | 63
    Grade 2 | 5 | 7 | 4 | 0 | 10 | 2 | 28
    Grade 3 | 1 | 0 | 0 | 0 | 5 | 1 | 7
    Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Missing | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to the Revised Response Criteria for Malignant Lymphoma (Parts A, B, and C)
Description: Objective response rate (ORR) per investigator was defined as the percentage of subjects with complete response (CR) or partial response (PR) through the end of study or prior to the start of new anti-cancer treatment (including stem cell transplant, and excluding consolidative radiotherapy) other than the study treatment. For Parts A, B, and C the response was assessed using the Revised Response Criteria for Malignant Lymphoma (Cheson 2007).
Time Frame: Up to 81 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A | Part B | Part C
Number analyzed (Participants) | 27 | 22 | 20
Percentage of participants | 93 [75.7 to 99.1] | 95 [77.2 to 99.9] | 85 [62.1 to 96.8]

2. Primary Outcome: ORR According to the Lugano Classification Revised Staging System for Nodal Non-Hodgkin and Hodgkin Lymphomas (Lugano Criteria) and the Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) (Part D)
Description: Objective response rate (ORR) per investigator was defined as the percentage of subjects with CR or PR through the end of study or prior to the start of new anti-cancer treatment (including stem cell transplant, and excluding consolidative radiotherapy) other than the study treatment. For Part D, the response was assessed using the Lugano Classification Revised Staging System for nodal non-Hodgkin and cHL (Lugano criteria) and the Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC).
Time Frame: Up to 60 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part D
Number analyzed (Participants) | 21
Percentage of participants | 86 [63.7 to 97.0]

3. Primary Outcome: ORR According to Modified Lugano Criteria Per Blinded Independent Central Review (BICR) (Parts E and F)
Description: Objective response rate (ORR) per investigator was defined as the percentage of subjects with CR or PR through the end of study or prior to the start of new anti-cancer treatment (including stem cell transplant, and excluding consolidative radiotherapy) other than the study treatment. For Parts E and F, the response was assessed per blinded independent central review (BICR) using the modified Lugano criteria.
Time Frame: Up to 31 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part E | Part F
Number analyzed (Participants) | 30 | 7
Percentage of participants | 60 [40.6 to 77.3] | 43 [9.9 to 81.6]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment-emergent AE (TEAE) is defined as a newly occurring or worsening AE after the first dose of any study drug component. Treatment-related AEs are defined as treatment-emergent AEs that are determined by the investigator to be related to the treatment on study. TEAEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.03). The CTCAE displays Grades 1 through 5, where Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences, Grade 5: Death related to AE.
Time Frame: Up to 122 months
Population: All subjects who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7
Participants
  Any TEAE | 27 | 22 | 20 | 21 | 30 | 7
  Treatment-related TEAE | 25 | 22 | 19 | 18 | 24 | 6
  Any grade 3 or higher TEAE | 17 | 10 | 18 | 16 | 18 | 7
  Treatment-related grade 3 or higher TEAE | 13 | 9 | 16 | 12 | 8 | 4
  Any treatment-emergent (TE) serious adverse event (SAE) | 5 | 4 | 13 | 4 | 14 | 4
  Treatment-related TE SAE | 3 | 3 | 9 | 0 | 3 | 1
  TEAE leading to treatment discontinuation | 11 | 11 | 12 | 5 | 9 | 3
  Treatment-related TEAE leading to treatment discontinuation | 11 | 9 | 8 | 2 | 5 | 2
  TEAE leading to death | 0 | 0 | 3 | 1 | 4 | 2
  Treatment-related TEAE leading to death | 0 | 0 | 0 | 0 | 1 | 1

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory values were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.03). The CTCAE displays Grades 1 through 5, where Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences, Grade 5: Death related to AE.
Time Frame: Up to 30 months
Population: All subjects who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7
Participants
  Hemoglobin High, Grade 1 | 2 | 1 | 0 | 1 | 1 | 0
  Hemoglobin High. Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin High. Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin High. Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Low, Grade 1 | 10 | 6 | 10 | 9 | 13 | 4
  Hemoglobin Low, Grade 2 | 5 | 6 | 6 | 5 | 6 | 1
  Hemoglobin Low, Grade 3 | 1 | 0 | 1 | 2 | 0 | 0
  Hemoglobin Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes Low, Grade 1 | 2 | 3 | 2 | 3 | 5 | 4
  Leukocytes Low, Grade 2 | 3 | 3 | 5 | 3 | 1 | 1
  Leukocytes Low, Grade 3 | 0 | 1 | 5 | 1 | 1 | 0
  Leukocytes Low, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocytes High, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes High, Grade 2 | 0 | 0 | 0 | 1 | 2 | 1
  Lymphocytes High, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Low, Grade 1 | 0 | 0 | 0 | 0 | 7 | 0
  Lymphocytes Low, Grade 2 | 4 | 7 | 2 | 6 | 7 | 2
  Lymphocytes Low, Grade 3 | 6 | 2 | 6 | 2 | 1 | 2
  Lymphocytes Low, Grade 4 | 0 | 0 | 9 | 1 | 0 | 0
  Neutrophils Low, Grade 1 | 0 | 0 | 0 | 2 | 0 | 0
  Neutrophils Low, Grade 2 | 3 | 4 | 5 | 2 | 2 | 1
  Neutrophils Low, Grade 3 | 2 | 1 | 3 | 2 | 2 | 2
  Neutrophils Low, Grade 4 | 0 | 2 | 1 | 1 | 1 | 0
  Platelets Low, Grade 1 | 4 | 2 | 8 | 3 | 5 | 2
  Platelets Low, Grade 2 | 2 | 1 | 2 | 1 | 0 | 0
  Platelets Low, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Low, Grade 4 | 0 | 0 | 0 | 1 | 0 | 0
  Alanine Aminotransferase High, Grade 1 | 8 | 9 | 6 | 16 | 7 | 0
  Alanine Aminotransferase High, Grade 2 | 4 | 1 | 0 | 0 | 0 | 0
  Alanine Aminotransferase High, Grade 3 | 1 | 0 | 0 | 2 | 0 | 0
  Alanine Aminotransferase High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin Low, Grade 1 | 8 | 6 | 9 | 9 | 6 | 3
  Albumin Low, Grade 2 | 3 | 3 | 5 | 6 | 4 | 0
  Albumin Low, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0
  Albumin Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase High, Grade 1 | 10 | 10 | 5 | 4 | 12 | 3
  Alkaline Phosphatase High, Grade 2 | 3 | 0 | 2 | 4 | 0 | 0
  Alkaline Phosphatase High, Grade 3 | 1 | 0 | 0 | 1 | 0 | 0
  Alkaline Phosphatase High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase High, Grade 1 | 0 | 0 | 0 | 5 | 0 | 0
  Amylase High, Grade 2 | 0 | 0 | 0 | 2 | 0 | 0
  Amylase High, Grade 3 | 0 | 0 | 0 | 3 | 0 | 0
  Amylase High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase High, Grade 1 | 14 | 8 | 8 | 16 | 9 | 0
  Aspartate Aminotransferase High, Grade 2 | 1 | 1 | 1 | 1 | 1 | 0
  Aspartate Aminotransferase High, Grade 3 | 2 | 0 | 0 | 1 | 1 | 0
  Aspartate Aminotransferase High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium Corrected for Albumin High, Grade 1 | 1 | 0 | 1 | 2 | 6 | 1
  Calcium Corrected for Albumin High, Grade 2 | 1 | 0 | 0 | 2 | 0 | 0
  Calcium Corrected for Albumin High, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium Corrected for Albumin High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium Corrected for Albumin Low, Grade 1 | 3 | 0 | 1 | 1 | 2 | 2
  Calcium Corrected for Albumin Low, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium Corrected for Albumin Low, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium Corrected for Albumin Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine High, Grade 1 | 20 | 14 | 12 | 12 | 18 | 3
  Creatinine High, Grade 2 | 2 | 1 | 2 | 2 | 1 | 0
  Creatinine High, Grade 3 | 0 | 1 | 0 | 1 | 0 | 0
  Creatinine High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Glomerular Filtration Rate, Estimated Low, Grade 1 | 0 | 0 | 0 | 0 | 2 | 1
  Glomerular Filtration Rate, Estimated Low, Grade 2 | 0 | 0 | 0 | 0 | 11 | 2
  Glomerular Filtration Rate, Estimated Low, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Glomerular Filtration Rate, Estimated Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose High, Grade 1 | 15 | 13 | 12 | 12 | 11 | 3
  Glucose High, Grade 2 | 10 | 6 | 3 | 5 | 8 | 2
  Glucose High, Grade 3 | 2 | 2 | 1 | 4 | 2 | 0
  Glucose High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose Low, Grade 1 | 0 | 1 | 0 | 1 | 1 | 0
  Glucose Low, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose Low, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase High, Grade 1 | 0 | 0 | 0 | 2 | 0 | 0
  Lipase High, Grade 2 | 0 | 0 | 1 | 2 | 0 | 0
  Lipase High, Grade 3 | 0 | 0 | 0 | 2 | 0 | 0
  Lipase High, Grade 4 | 0 | 0 | 0 | 2 | 0 | 0
  Phosphate Low, Grade 1 | 9 | 8 | 2 | 7 | 0 | 0
  Phosphate Low, Grade 2 | 2 | 5 | 3 | 6 | 4 | 0
  Phosphate Low, Grade 3 | 2 | 0 | 4 | 2 | 0 | 0
  Phosphate Low, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium High, Grade 1 | 1 | 1 | 0 | 0 | 1 | 0
  Potassium High, Grade 2 | 0 | 0 | 0 | 1 | 0 | 0
  Potassium High, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium High, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium Low, Grade 1 | 6 | 5 | 5 | 8 | 1 | 2
  Potassium Low, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium Low, Grade 3 | 2 | 0 | 3 | 1 | 2 | 0
  Potassium Low, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0
  Sodium High, Grade 1 | 0 | 2 | 2 | 0 | 0 | 0
  Sodium High, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium High, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium Low, Grade 1 | 11 | 7 | 4 | 9 | 7 | 0
  Sodium Low, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium Low, Grade 3 | 1 | 1 | 3 | 3 | 0 | 1
  Sodium Low, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0
  Total Bilirubin High, Grade 1 | 3 | 2 | 4 | 3 | 2 | 0
  Total Bilirubin High, Grade 2 | 0 | 0 | 1 | 4 | 0 | 0
  Total Bilirubin High, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0
  Total Bilirubin High, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Urate High, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urate High, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Urate High, Grade 3 | 5 | 7 | 4 | 9 | 4 | 0
  Urate High, Grade 4 | 3 | 0 | 0 | 2 | 0 | 0

6. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the percentage of patients with CR
Time Frame: Up to 81 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7
Percentage of participants | 70 [49.8 to 86.2] | 64 [40.7 to 82.8] | 75 [50.9 to 91.3] | 67 [43.0 to 85.4] | 30 [14.7 to 49.4] | 43 [9.9 to 81.6]

7. Secondary Outcome: Duration of Complete Response
Description: Duration of CR per investigator was defined as the time from start of the first documentation of CR to the first documentation of tumor progression or to death due to any cause, whichever came first. For Parts E and F, the assessment was per BICR.
Time Frame: Up to 81 months
Population: All subjects with CR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 19 | 14 | 15 | 14 | 10 | 2
Months | 7.4 [5.1 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | NA [14.7 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | NA [2.8 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | NA [6.6 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | NA [7.4 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | NA [NA to NA] — Follow-up duration too short relative to event accumulation to estimate median, upper limit, and lower limit.

8. Secondary Outcome: Duration of Objective Response
Description: Duration of response per investigator was defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression (PD) based on radiographic evidence of progression or to death due to any cause, whichever came first. For Parts E and F, the assessment was per BICR.
Time Frame: Up to 81 months
Population: All subjects with CR/PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 25 | 21 | 17 | 18 | 18 | 3
Months | 7.6 [5.1 to 67.7] | 46.0 [8.5 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | NA [3.6 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | NA [12.7 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | 7.4 [7.4 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | NA [11.3 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit.

9. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) per investigator was defined as the time from start of study treatment to first documentation of tumor progression or to death due to any cause, whichever came first. For Parts E and F, the assessment was per BICR.
Time Frame: Up to 83 months
Population: All subjects who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7
Months | 8.6 [6.3 to 40.1] | 47.2 [10.8 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | 32.5 [4.0 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | NA [9.4 to NA] — Follow-up duration too short relative to event accumulation to estimate median and upper limit. | 8.7 [5.1 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | 10.5 [0.5 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit.

10. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) per investigator was defined as the percentage of subjects with CR, PR, or SD, per investigator assessment of best clinical response per Cheson 2007. For Parts E and F, the assessment was per BICR.
Time Frame: Up to 81 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 27 | 22 | 20 | 21 | 30 | 7
Percentage of participants | 100 [87.2 to 100.0] | 95 [77.2 to 99.9] | 85 [62.1 to 96.8] | 90 [69.6 to 98.8] | 77 [57.7 to 90.1] | 57 [18.4 to 90.1]

11. Secondary Outcome: ORR According to Lugano Criteria Per BICR (Parts E and F)
Description: Objective response rate (ORR) per investigator was defined as the percentage of subjects with CR or PR through the end of study or prior to the start of new anti-cancer treatment (including stem cell transplant, and excluding consolidative radiotherapy) other than the study treatment.
Time Frame: Up to 31 months
Population: All subjects who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part E | Part F
Number analyzed (Participants) | 30 | 7
Percentage of participants | 67 [47.2 to 82.7] | 43 [9.9 to 81.6]

12. Secondary Outcome: B Symptom Resolution Rate
Description: B symptom resolution rate per investigator was defined as the percentage of subjects with lymphoma-related B symptoms at baseline who achieved resolution of all B symptoms at any time during the treatment period.
Time Frame: Up to 42 weeks
Population: Subjects with any B symptom at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 9 | 2
Percentage of participants | 100 [47.8 to 100.0] | 100 [54.1 to 100.0] | 86 [42.1 to 99.6] | 67 [22.3 to 95.7] | 0 [NA to NA] — No participants achieved B symptom resolution | 0 [NA to NA] — No participants achieved B symptom resolution

13. Secondary Outcome: Number of Participants With Brentuximab Vedotin Antitherapeutic Antibodies (ATA)
Time Frame: Up to 30 months
Population: Subjects with a baseline and at least one post-baseline sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
Number analyzed (Participants) | 26 | 22 | 17 | 18 | 26 | 6
Participants
  Baseline Negative | 23 | 20 | 16 | 17 | 24 | 6
  Baseline Negative - Negative post-baseline | 14 | 12 | 5 | 12 | 17 | 6
  Baseline Negative - Positive post-baseline | 9 | 8 | 11 | 5 | 7 | 0
  Baseline Positive | 3 | 2 | 1 | 1 | 2 | 0
  Baseline Positive - Negative post-baseline | 3 | 2 | 1 | 1 | 2 | 0
  Baseline Positive: Treatment-boosted post-baseline | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Nivolumab Antitherapeutic Antibodies (ATA) (Part D Only)
Time Frame: Up to 30 months
Population: Subject with baseline negative anti-drug antibody (ADA)
Measure: Count of Participants; unit: Participants
Arm/Group | Part D
Number analyzed (Participants) | 17
Participants
  Cycle 1 (Pre-dose nivolumab) | 0
  First Positive Cycle (pre-dose) - Cycle 2 | 4
  First Positive Cycle (pre-dose) - Cycle 8 | 1
  Any positive post-baseline | 5

15. Secondary Outcome: Overall Survival (Parts E and F Only)
Description: Overall survival (OS) per investigator was defined as the time from date of enrollment to date of death due to any cause.
Time Frame: Up to 44 months
Population: All subjects who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part E | Part F
Number analyzed (Participants) | 30 | 7
Months | 31.8 [14.8 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit. | 12.6 [0.5 to NA] — Follow-up duration too short relative to event accumulation to estimate upper limit.

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events, Serious Adverse Events, and All-Cause Mortality were followed for up to 122 months
Description: The population for all-cause mortality and adverse events includes participants who received at least one dose of study drug.
Arm/Group | Part A | Part B | Part C | Part D | Part E | Part F
All-Cause Mortality (participants affected / at risk) | 13/27 | 9/22 | 12/20 | 4/21 | 10/30 | 5/7
Serious Adverse Events (participants affected / at risk) | 5/27 | 4/22 | 13/20 | 4/21 | 14/30 | 4/7
Other Adverse Events (participants affected / at risk) | 27/27 | 22/22 | 20/20 | 21/21 | 27/30 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=27) | Part B (N=22) | Part C (N=20) | Part D (N=21) | Part E (N=30) | Part F (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=27) | Part B (N=22) | Part C (N=20) | Part D (N=21) | Part E (N=30) | Part F (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (5) | 3 (4) | 2 (2) | 1 (1) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (5) | 5 (7) | 1 (4) | 1 (1) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (6) | 3 (3) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (9) | 10 (12) | 7 (7) | 10 (11) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 6 (9) | 17 (21) | 9 (10) | 7 (12) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 9 (11) | 13 (16) | 8 (8) | 10 (12) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (4) | 4 (5) | 2 (2) | 4 (4) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (3) | 3 (3) | 7 (11) | 2 (2) | 0 (0)
Fatigue (General disorders) | 12 (12) | 10 (10) | 10 (11) | 16 (22) | 9 (11) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 7 (8) | 6 (7) | 5 (5) | 3 (4) | 4 (4) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 4 (5) | 7 (8) | 7 (11) | 2 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6) | 3 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (6) | 5 (11) | 2 (2) | 1 (1) | 2 (3)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 5 (5) | 5 (5) | 4 (5) | 4 (4) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 5 (5) | 9 (9) | 7 (7) | 8 (9) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 7 (8) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 5 (8) | 3 (5) | 2 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (8) | 1 (1) | 7 (10) | 5 (5) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 1 (1) | 2 (4) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (4) | 4 (8) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 3 (3) | 5 (5) | 4 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (7) | 1 (1) | 4 (5) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 5 (5) | 2 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (22) | 17 (21) | 8 (8) | 10 (16) | 14 (16) | 4 (8)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4) | 4 (5) | 3 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (14) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 5 (5) | 3 (3) | 6 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (6) | 4 (4) | 3 (6) | 6 (10) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (10) | 5 (7) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 6 (6) | 6 (11) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT01716806/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT01716806/SAP_001.pdf